CLINICAL TRIAL: NCT04529135
Title: The Effect of Dexmedetomidine During Opioid Free Anesthesia on Postoperative Recovery After Gastrectomy : A Randomized Controlled Trial
Brief Title: The Effect of Dexmedetomidine During Opioid Free Anesthesia on Postoperative Recovery After Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Ji-young Kim, Associate professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-0219-002
Record Dates: First submitted 2020-08-11; First posted 2020-08-27 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Dexmedetomidine; Remifentanil

STUDY DESIGN:
Intervention Model Description: Randomized Double-blind Controlled Study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients are divided into the Dexmedetomidine group / control group by random assignment. Using a table of computer-generated random numbers(s), assign 68 people to each county by 34 people. Random tables, in turn, seal the results in an opaque envelope. An anesthesiologist who is unaware of the content of this study and does not participate in the study receives information only about drug administration and is in charge of anesthesia, and does not disclose information about the assigned group to postoperative observers. Also, they don't disclose information about the assigned group to the surgeon.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): IV,0.2~0.8 µg/kg/hr
  Interventions: Drug: Dexmedetomidine
- Remifentanil (Active Comparator): IV,0.05~0.2 µg/kg/min
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Dexmedetomidine — The prepared drug marks the assigned group as unknown. In both groups, the test drug marked as unknown begins to be administered in an anesthetic induction. When the patient arrives in the operating room, electrocardiogram, noninvasive blood pressure, and bispectral index (BIS) monitoring is performed. In both groups, 2 mg/kg of propofol induces general anesthesia, intubates after administration of rocuronium 0.6 mg/kg, and maintains anesthesia with sevoflurane 1.5-2.5 vol%. Use 0.075 mg of palonosetrone as an antiemetics after inducing anesthesia. Adjust the inhalation anesthetic to maintain BIS 40-60 , mechanical ventilation to maintain the Tidal volume of 8 ml/kg, PEEP 5 mmHg and end-tidal carbon dioxide (EtCO2) of 35-40 mmHg. Push 1mcg of fentanyl and 1g of acetaminophen per kg for pain control 20 minutes before the end of surgery.
  Arms: Dexmedetomidine
Drug: Remifentanil — The prepared drug marks the assigned group as unknown. In both groups, the test drug marked as unknown begins to be administered in an anesthetic induction. When the patient arrives in the operating room, electrocardiogram, noninvasive blood pressure, and bispectral index (BIS) monitoring is performed. In both groups, 2 mg/kg of propofol induces general anesthesia, intubates after administration of rocuronium 0.6 mg/kg, and maintains anesthesia with sevoflurane 1.5-2.5 vol%. Use 0.075 mg of palonosetrone as an antiemetics after inducing anesthesia. Adjust the inhalation anesthetic to maintain BIS 40-60 , mechanical ventilation to maintain the Tidal volume of 8 ml/kg, PEEP 5 mmHg and end-tidal carbon dioxide (EtCO2) of 35-40 mmHg. Push 1mcg of fentanyl and 1g of acetaminophen per kg for pain control 20 minutes before the end of surgery.
  Arms: Remifentanil

SUMMARY:
"Want to know the effect of dexmedetomidine during opioid free anesthesia on postoperative recovery after gastrectomy. Patients undergoing open gastrectomy are divided into dexmedetomidine group and control(remifentanil) group, administered during surgery, and compared with the speed of postoperative intestinal function recovery. Based on our institution's previous record, the average recovery time was 6 ± 1.4 days. Given that it is clinically significant to reduce recovery time by 20%, Alpha 0.05 and Power 80% require 31 samples per group, and assuming a 10% dropout rate, the total number of samples needed is 68.Subjects are patients aged 19 to 75 who are subject to open gastretomy planned by a gastric cancer. The exclusion criteria include American Society of Anesthesiology grade 3 or higher, patients who have previously been treated for cancer, patients with cancer other than the stomach, patients with drug allergies, weight less than 60kg, BMI > 30 kg/m2, patients who are unable to communicate and are unable to read consent (e.g., illiteracy, foreigners, etc.). The research method is a Randomized double-blind controlled study, and the assignment of both drugs is unknown and is used to maintain anesthesia in the form of continuous injection during surgery. Primary outcome is the recovery period satisfying the following. 1)intestinal gas passage 2) tolerance of soft bland diet (SBD) for 24 hr. 3) safe ambulation without assistance 4) no requirement iv analgesics after discontinuation of PCA (VAS <4). 5) no abnormal physical signs or laboratory test. The secondary outcomes are maximum VAS, post-operative hospital stay, complications and readmission rate at 3 months F/U time, post-operative period analgesic requirement, incidence of opioid related side effect.

ELIGIBILITY:
Inclusion Criteria:

-patients undergoing open gastrectomy for gastric cancer

Exclusion Criteria:

* American Society of Anesthesiology grade 3 or higher
* history of chemotherapy
* diagosis of cancer in other organs
* history of drug allergy
* weight less than 60kg
* BMI over 30 kg/m2 patient
* cognitive impairment
* gait disturbance

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
postoperative recovery time | 3 months
  number of days satisfying all following criteria 1)intestinal gas passage 2) tolerance of soft bland diet (SBD) for 24 hr. 3) safe ambulation without assistance 4) no requirement iv analgesics after discontinuation of PCA (VAS <4). 5) no abnormal physical signs or laboratory test.

SECONDARY OUTCOMES:
maximum pain score | 3 months
  Visual analogue scale (VAS: 0-10)
post-operative hospital stay | 3 months
  days
complications and readmission rate at 3 months F/U time | 3 months
  incidence
post-operative period analgesic requirement | 3 months
  number of analgesic requirement despite intravenous patient controlled analgesia
opioid related side effect. | 3 months
  incidence of nausea, vomiting and pruritus

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea